CLINICAL TRIAL: NCT05314153
Title: Open Label Study of the Efficacy, Safety and Tolerability of Zulresso in the Treatment of Adult Women With Postpartum Psychosis
Brief Title: Effects Zulresso on Postpartum Psychosis
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: University of North Carolina, Chapel Hill (Other)
Collaborators: Sage Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 20-0812
Record Dates: First submitted 2022-03-28; First posted 2022-04-06 (Actual); Last update posted 2024-08-26 (Actual); Status verified 2024-04

CONDITIONS: Postpartum Psychosis
MeSH Terms: interventions — brexanolone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Open Label - Active Drug (Experimental): Brexanolone (zulresso) infusion arm. All patients enrolled will receive active treatment with brexanolone.
  Interventions: Drug: Brexanolone

INTERVENTIONS:
Drug: Brexanolone — Brexanolone injection is an Federal Drug Administration (FDA)-approved drug to treat postpartum depression. It is administered via continuous intravenous infusion over a 60-hour time period.
  Other Names: Zulresso

SUMMARY:
This is an open-label, proof of concept trial to investigate the efficacy, safety and tolerability of Zulresso (brexanolone) administered to adult female subjects diagnosed with postpartum psychosis. This study will provide critical pilot data to determine whether there is similar treatment efficacy among patients with postpartum psychosis as observed to date in patients with postpartum depression.

DETAILED DESCRIPTION:
This is a single site, open label study design to evaluate the efficacy, safety and tolerability of Zulresso in female subjects diagnosed with postpartum psychosis.

Participants will be consented, and if possible, participation will be discussed with available family members. Participants will take a consent questionnaire prior to consenting to ensure the voluntary nature and understanding of study procedures. Participants will undergo a screening visit including diagnostic interviews, clinical laboratory assessments and an EKG to determine eligibility. If eligible, participants will be admitted in-patient to UNC Hospitals and administered a continuous 60-hour infusion of Zulresso using the approved FDA REMS protocol for postpartum depression. A target dose of 90 μg/kg/hour will be administered over a period of 2.5 days following a strict tapering schedule. Monitoring will occur for an additional 12 hours after the infusion. The subject will participate in 6 follow up visits at day 7 post-infusion, day 14, day 21, day 30, day 60 and day 90.

ELIGIBILITY:
Inclusion Criteria:

* All participating subjects sign an informed consent form;
* Age 18-45 years old;
* Onset of affective psychosis or mania symptoms in the 3rd trimester, within 4 weeks of delivery, or within 4 weeks of weaning;
* Clinician diagnosis of affective psychosis or mania;
* ≤12 months postpartum at screening

Exclusion Criteria:

* Positive pregnancy test at screening or day 1;
* Recent pregnancy did not result in a live birth;
* Subject is in renal failure;
* Subject is in hepatic failure;
* Subject is anemic (hemoglobin ≤10 g/dL);
* Untreated or inadequately treated hypothyroidism or hyperthyroidism;
* History of schizophrenia, and/or schizoaffective disorder;
* Current/active alcohol or drug abuse

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 10 (Actual)
Dates: Start 2022-02-23 (Actual); Primary Completion 2024-06-01 (Actual); Study Completion 2024-06-01 (Actual)

PRIMARY OUTCOMES:
Change in Positive and Negative Syndrome Scale (PANSS) score | Baseline to post-treatment day 7
  The PANSS is a standardized, clinical interview that rates the presence and severity of psychosis. The PANSS yields a total average symptom score, based on 30 items rated from one to seven (range=30-210). Higher scores indicate more severe symptoms.
Change in Young Mania Rating Scale (YMRS) score | Baseline to post-treatment day 7
  The Young Mania Rating Scale (YMRS) is one of the most frequently utilized rating scales to assess manic symptoms. The scale has 11 items and is based on the patient's subjective report of his or her clinical condition over the previous 48 hours. The items are selected based upon the core symptoms of mania. The YMRS total score ranges from 0 to 60 where higher scores indicate more severe symptoms.

SECONDARY OUTCOMES:
Change in Hamilton Rating Scale for Depression (HAM-D) | Baseline to post-treatment day 7
  The 17-item HAM-D will be used to rate the severity of depression in subjects who are already diagnosed as depressed. The HAM-D comprises individual ratings related to the following symptoms: depressed mood (sadness, hopeless, helpless, worthless), feelings of guilt, suicide, insomnia (early, middle, late), work and activities, retardation (slowness of thought and speech; impaired ability to concentrate; decreased motor activity), agitation, anxiety (psychic and somatic), somatic symptoms (gastrointestinal and general), genital symptoms, hypochondriasis, loss of weight, and insight. The HAM-D maximum score is 52 for the 17 items with a higher score indicating more severe symptoms.
Change in Edinburgh Postnatal Depression Scale (EPDS) | Baseline to post-treatment day 7
  The EPDS is a 10-item subject-rated depressive symptom severity scale specific to the perinatal period. The EPDS maximum score is 30 with higher scores indicating more severe symptoms.
Change in Clinical Global Impression Scale (CGI) | Baseline to post-treatment day 7
  The CGI is a validated scale to allow clinicians to measure a subject's change in illness severity from baseline. The CGI scale consists of three items. Only the first two items (CGI-S and CGI-I) will be used in this study. The CGI-S uses a seven-point Likert scale to rate the severity of the subject's illness at the time of assessment, relative to the clinician's past experience with subjects who have the same diagnosis. The CGI-I employs a seven-point Likert scale to measure the overall improvement in the subject's condition post-treatment. The CGI-S is rated on a 7-point scale, with the severity of illness scale using a range of responses from 1 (normal) through to 7 (amongst the most severely ill patients). CGI-I scores range from 1 (very much improved) through to 7 (very much worse).

CONTACTS AND LOCATIONS:
Overall Officials: Samantha Meltzer-Brody, MD, MPH, Principal Investigator — University of North Carolina, Chapel Hill
Locations (1):
- UNC Hospitals, Chapel Hill, North Carolina, United States

IPD SHARING:
Plan to Share IPD: Yes
Deidentified individual data that supports the results will be shared beginning 9 to 36 months following publication provided the investigator who proposes to use the data has approval from an Institutional Review Board (IRB), Independent Ethics Committee (IEC), or Research Ethics Board (REB), as applicable, and executes a data use/sharing agreement with UNC.
Supporting Information: Study Protocol, SAP
Time Frame: Data will be available by investigator request starting 9 months following publication and continue through 36 months afterwards.
Access Criteria: Investigator has approved IRB, IEC, or REB and an executed data use/sharing agreement with UNC.

REFERENCES:
- [Background] Kanes S, Colquhoun H, Gunduz-Bruce H, Raines S, Arnold R, Schacterle A, Doherty J, Epperson CN, Deligiannidis KM, Riesenberg R, Hoffmann E, Rubinow D, Jonas J, Paul S, Meltzer-Brody S. Brexanolone (SAGE-547 injection) in post-partum depression: a randomised controlled trial. Lancet. 2017 Jul 29;390(10093):480-489. doi: 10.1016/S0140-6736(17)31264-3. Epub 2017 Jun 12. PMID 28619476
- [Background] Meltzer-Brody S, Colquhoun H, Riesenberg R, Epperson CN, Deligiannidis KM, Rubinow DR, Li H, Sankoh AJ, Clemson C, Schacterle A, Jonas J, Kanes S. Brexanolone injection in post-partum depression: two multicentre, double-blind, randomised, placebo-controlled, phase 3 trials. Lancet. 2018 Sep 22;392(10152):1058-1070. doi: 10.1016/S0140-6736(18)31551-4. Epub 2018 Aug 31. Erratum In: Lancet. 2018 Sep 29;392(10153):1116. doi: 10.1016/S0140-6736(18)32288-8. PMID 30177236
- [Background] Kanes SJ, Colquhoun H, Doherty J, Raines S, Hoffmann E, Rubinow DR, Meltzer-Brody S. Open-label, proof-of-concept study of brexanolone in the treatment of severe postpartum depression. Hum Psychopharmacol. 2017 Mar;32(2):e2576. doi: 10.1002/hup.2576. PMID 28370307
- [Background] Scott LJ. Brexanolone: First Global Approval. Drugs. 2019 May;79(7):779-783. doi: 10.1007/s40265-019-01121-0. PMID 31006078